CLINICAL TRIAL: NCT03334305
Title: ACTION Trial: Adoptive Cellular Therapy Following Dose-Intensified Temozolomide in Newly-diagnosed Pediatric High-grade Gliomas (Phase I).
Brief Title: Adoptive Cellular Therapy in Pediatric Patients With High-grade Gliomas
Acronym: ACTION
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: due to lack of accrual/feasibility to complete accrual due to competing trials
Sponsor: University of Florida (Other)
Collaborators: National Pediatric Cancer Foundation (Other); National Cancer Institute (NCI) (NIH); Moffitt Clinical Research Network (MCRN) (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB201701867-N; R01CA195563 (NIH); OCR15852 (Other: Universiy of Florida)
Record Dates: First submitted 2017-10-26; First posted 2017-11-07 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Malignant Glioma; High Grade Glioma
Keywords: Immunotherapy; Pediatric; Vaccine Therapy; Young adult; Immune system; Dendritic Cell
MeSH Terms: conditions — Glioma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Diphtheria-Tetanus Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Dose-intensified TMZ with TTRNA-DC vaccines with GM-CSF and TTRNA-xALT plus Td vaccine without Autologous Hematopoietic Stem cells (HSCs)
  Interventions: Biological: TTRNA-DC vaccines with GM-CSF; Drug: Dose-intensified TMZ; Biological: TTRNA-xALT; Drug: Td vaccine
- Group B (Experimental): Dose-intensified TMZ with TTRNA-DC vaccines with GM-CSF and TTRNA-xALT plus Td vaccine with Autologous Hematopoietic Stem cells (HSCs)
  Interventions: Biological: TTRNA-DC vaccines with GM-CSF; Drug: Dose-intensified TMZ; Biological: Autologous Hematopoietic Stem cells (HSCs); Biological: TTRNA-xALT; Drug: Td vaccine

INTERVENTIONS:
Biological: TTRNA-DC vaccines with GM-CSF — After chemoradiation subjects will receive the first cycle of dose-intensified TMZ followed by three biweekly TTRNA-DC vaccines with GM-CSF. Monthly DC vaccines will be given during TMZ Cycles 2-5 for Groups A and B and 48-96 hours after completion of TMZ Cycle 6 Day 21 for Group A and 12-36 hours after HSCs for Group B. All subjects will receive an additional two bi-weekly vaccines during Cycle 6 for a total of 10 DC vaccines. All DC vaccines will be embedded with GM-CSF (150 µg per injection) and given intradermal.
Drug: Dose-intensified TMZ — After chemoradiation, subjects will receive the first cycle of dose-intensified TMZ followed by three biweekly TTRNA-DC vaccines with GM-CSF. All subjects will have an additional five cycles of dose-intensified TMZ (for a total of 6 Cycles) with concurrent monthly DC vaccinations.
Biological: Autologous Hematopoietic Stem cells (HSCs) — Prior to chemoradiation, enrolled subjects will undergo a mobilized leukapheresis for collection of PBSCs and PBMCs for generation of DCs. One group will receive recommended dose of > 2 x 106 CD34+ HSCs/kg. Subjects enrolled in Group B will receive HSCs during TMZ Cycle 6 before receiving DC vaccine and T-cell infusion.
  Arms: Group B
Biological: TTRNA-xALT — During TMZ Cycle 6 and with DC vaccine #8, an infusion of T-cells will be administered to all subjects.
Drug: Td vaccine — A full Td booster vaccine will be administered IM at Vaccine #1 to all subjects, and vaccine site pretreatment will be administered to all subjects prior to Vaccine#3, #6, and #8.

SUMMARY:
It is believed that the body's immune system protects the body by attacking and killing tumor cells. T-lymphocytes (T-cells) are part of the immune system and can attack when they recognize special proteins on the surface of tumors. In most patients with advanced cancer, T-cells are not stimulated enough to kill the tumor. In this research study, we will use a patient's tumor to make a vaccine which we hope will stimulate T-cells to kill tumor cells and leave normal cells alone.

High grade gliomas (HGGs) are very aggressive and difficult for the body's immune system to attack. Before T-cells can become active against tumor cells, they require strong stimulation by special "stimulator" cells in the body called Dendritic Cells (DCs) which are also part of the immune system. DCs can recognize the cancer cells and then activate the T lymphocytes, and create this strong stimulation.

The purpose of this research study is to learn whether anti-tumor T-cells and anti-tumor DC vaccines can be given safely. Most importantly, this study is also to determine whether the T-cells and DC vaccines can stimulate a person's immune system to fight off the tumor cells in the brain.

DETAILED DESCRIPTION:
It is believed that the body's immune system protects the body by attacking and killing tumor cells. T-lymphocytes (T-cells) are part of the immune system and can attack when they recognize special proteins on the surface of tumors. But in most patients with advanced cancer, T-cells are not stimulated enough to kill the tumor. In this research study, we will use your tumor to make a vaccine which we hope will stimulate your T-cells to kill tumor cells and leave your normal cells alone.

High grade gliomas (HGGs) are very aggressive and difficult for the body's immune system to attack. Before T-cells can become active against tumor cells, they require strong stimulation by special "stimulator" cells in the body called Dendritic Cells (DCs) which are also part of the immune system. DCs can recognize the cancer cells and then activate the T lymphocytes, and create this strong stimulation.

The purpose of this research study is to learn whether anti-tumor T-cells and anti-tumor DC vaccines can be given safely. Most importantly, this study is also to determine whether the T-cells and DC vaccines can stimulate your immune system to fight off the tumor cells in your brain. When the vaccine for this study is made, dendritic cells will be loaded with genetic material called RNA (ribonucleic acid) from your tumor to stimulate the dendritic cells. The vaccine has two components given at different times after chemoradiation and throughout chemotherapy cycles. The first part, the DC vaccine, involves RNA loaded dendritic cells that are given under the skin at several time points in the study and the second part, xALT vaccine, is a single infusion of tumor-specific T cells delivered through one of two peripheral IV catheters that are placed prior to infusion. This vaccine is investigational which means that it is not approved by the US Food and Drug Administration (FDA) and is being tested in research studies.

It is hoped that by injecting the DC vaccine into your skin and infusing the T-cells into your blood, your immune system will be activated against the tumor. Once it is activated against the tumor, your immune system may recognize and attack the tumor cells in your brain and not attack normal cells. Use of a vaccine that stimulates your immune system is called immunotherapy.

ELIGIBILITY:
Screening Eligibility:

* Patients with histologically confirmed WHO Grade III or IV malignant glioma
* Scheduled for definitive surgical resection of suspected HGG (biopsy only subjects are not eligible for this study)

Post-Surgical Resection Eligibility

* Histologically confirmed WHO Grade III or IV malignant glioma
* Karnofsky Performance Status (KPS) of ≥ 60% (KPS for ≥ 16 years of age) or Lansky performance Score (LPS) of ≥ 60 (LPS for < 16 years of age) assessed within 2 weeks prior to registration
* Bone Marrow: ANC (Absolute neutrophil count) ≥ 1000/µl (unsupported); Platelets ≥ 100,000/µl (unsupported for at least 3 days); Hemoglobin > 8 g/dL (may be supported)
* Renal:Serum creatinine ≤ upper limit of institutional normal
* Hepatic: Bilirubin ≤ 1.5 times upper limit of institutional normal for age. SGPT (ALT) ≤ 3 times upper limit of institutional normal for age. SGOT (AST) ≤ 3 times upper limit of institutional normal for age.
* Signed informed consent according to institutional guidelines.
* Patient or patient guardian consent to PBSC harvest following registration.
* Subjects of childbearing or child-fathering potential must be willing to use medically acceptable forms of birth control while being treated on this study.
* Subjects with post-surgical neurological deficits should have deficits that are stable for a minimum of 1 week prior to leukapheresis.

Exclusion Criteria:

* Pregnant or need to breast feed during the study period (Negative serum pregnancy test required).
* Known autoimmune or immunosuppressive disease or human immunodeficiency virus infection.
* Subjects with significant renal, cardiac (congestive cardiac failure, myocardial infarction, myocarditis), pulmonary, hepatic or other organ dysfunction.
* Severe or unstable concurrent medical conditions.
* Prior allergic reaction to TMZ, GM-CSF, or Td
* Subjects who are unwilling or unable to receive treatment and undergo follow-up evaluations at the enrolled Sunshine Project Consortium treatment site.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Evaluate safety of TTRNA-DCs and TTRNA-xALT | From first DC Vaccine through 30 days after administration of the last dose of trial drug or subject death
  Percentage of subjects with grade 3 or greater adverse events

SECONDARY OUTCOMES:
Determine feasibility of completing treatment | Up to 10 months
  Number of subjects completing treatment
Anti-tumor immune responses | up to 10 months
  Estimate the mean difference and the variation in INF gamma secretion
Progression-free survival (PFS) | Up to 8 years
  Median time to progression
Overall survival (OS) | Up to 8 years
  Median time to death

CONTACTS AND LOCATIONS:
Overall Officials: Elias Sayour, MD, PhD, Principal Investigator — University of Florida; Duane Mitchell, MD, PhD, Study Chair — University of Florida
Locations (3):
- United States (3):
  - Children's of Alabama at UAB, Birmingham, Alabama
  - Children's National Hospital, Washington D.C., District of Columbia
  - UF Health Shands Children's Hospital, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT03334305/ICF_000.pdf